CLINICAL TRIAL: NCT01926509
Title: A 28-Day Multiple-Dose Titration Study to Assess the Effects of MK-8892 on Safety, Tolerability and Pharmacokinetics in Subjects With Pulmonary Arterial Hypertension
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of MK-8892 in Participants With Pulmonary Arterial Hypertension (PAH) (MK-8892-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8892-005; 2013-002529-51 (EudraCT Number); MK-8892-005 (Other: Merck)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-8892 Panel A (Experimental): Participants will be administered MK-8892 once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 3 mg (Days 15-21), 4 mg (Days 22-28).
  Interventions: Drug: MK-8892
- MK-8892 Panel B (Experimental): Participants will be administered MK-8892 orally, once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 4 mg (Days 15-21), 4 mg (Days 22-28).
  Interventions: Drug: MK-8892
- MK-8892 Panel C (Experimental): Participants will be administered MK-8892 orally, once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 4 mg (Days 15-21), up to 8 mg (Days 22-28).
  Interventions: Drug: MK-8892
- Placebo (Panels A and B) (Placebo Comparator): Participants will be administered placebo to MK-8892 once daily for 28 days.
  Interventions: Drug: Placebo for MK-8892

INTERVENTIONS:
Drug: MK-8892
  Arms: MK-8892 Panel A; MK-8892 Panel B; MK-8892 Panel C
Drug: Placebo for MK-8892
  Arms: Placebo (Panels A and B)

SUMMARY:
This study will evaluate the safety, tolerability, and PK of MK-8892 in participants with pulmonary arterial hypertension. The primary hypothesis is that the geometric mean of MK-8892 area under the concentration time-curve from Hour 0 to 24 hours (AUC0-24hr) in participants with PAH, will be equal to or greater than the efficacious exposure in humans of 0.6 μM•hr.

ELIGIBILITY:
Inclusion Criteria:

* If female, cannot be pregnant or breastfeeding. Females of reproductive potential must agree to agree to use (and/or have their partner use) two (2) acceptable methods of birth control throughout the study and until 2 weeks after the last dose of study drug is administered
* Body mass index (BMI) ≤34 kg/m^2 and a total body weight >40 kg (>88 lbs)
* Has Group 1 pulmonary hypertension (PAH) as defined by the Dana Point 2008 Clinical Classification including: idiopathic PAH (IPAH), Heritable PAH, Drug and toxin-induced PAH, PAH associated with connective tissue disease or congenital heart disease (repaired simple cardiac defects at least 1 year status post corrective surgery, with no residual intracardiac or extracardiac shunt)
* On a stable regimen of background therapy for at least 3 months prior to starting study drug
* Have history of right heart catheterization within two years demonstrating pulmonary arterial hypertension
* Had pulmonary function testing within one year of starting study medication demonstrating total lung capacity (TLC) >70% predicted, forced expiratory volume in 1 second (FEV1) >70% predicted
* Have hemoglobin >75% of the lower limit of the normal range

Exclusion Criteria:

* Pulmonary hypertension subtypes including the following according to Dana Point 2008 Clinical Classification: human immunodeficiency virus (HIV) infection, portal hypertension, schistosomiasis, chronic hemolytic anemia, persistent pulmonary hypertension of the newborn (PPHN), pulmonary hypertension due to left heart diseases such as systolic dysfunction, diastolic dysfunction or valvular disease, pulmonary hypertension due to lung diseases and/or hypoxia (e.g. chronic obstructive pulmonary disease, interstitial lung disease, other pulmonary diseases with mixed restrictive and obstructive pattern, sleep-disordered breathing, alveolar hypoventilation disorders, chronic exposure to high altitude, and developmental abnormalities), chronic thromboembolic pulmonary hypertension (CTEPH), hematologic disorder (myeloproliferative disorders, splenectomy), systemic disorders (sarcoidosis, pulmonary Langerhans cell histiocytosis, lymphangioleiomyomatosis, neurofibromatosis, vasculitis), metabolic disorders (glycogen storage disease, Gaucher disease, thyroid disorders) or other disorder (tumoral obstruction, fibrosing mediastinitis, chronic renal failure on dialysis)
* Have secondary forms of pulmonary hypertension due to pulmonary veno-occlusive disease (PVOD), or pulmonary capillary hemangiomatosis (PCH)
* Resting systolic blood pressure <105 mmHg, or resting heart rate ≥110/min
* Family history of Long QT Syndrome
* Uncorrected hypokalemia or hypomagnesemia
* Taking medications that are potent inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4) including but not limited to cyclosporine, systemic itraconazole or ketoconazole, glyburide, erythromycin, clarithromycin, or telithromycin, nefazodone, protease inhibitors, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifampicin, St John's wort, diltiazem and verapamil) or has discontinued treatment <3 weeks prior to the start of the study. Concomitant medications, including anticoagulants, angiotensin converting enzyme (ACE) -inhibitors, diuretics, bosentan, ambrisentan and selected calcium channel blockers (e.g., amlodipine) may be allowed at the discretion of the investigator with the concurrence of the Sponsor.
* Unable to refrain from or anticipates the use of organic nitrates (e.g. nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, pentaerythritol) beginning approximately 2 weeks before start of study and throughout the study
* Unable to refrain from or anticipates the use of prostanoid therapies beginning approximately 2 weeks before start of study and throughout the study
* Consume excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Major surgery or donated blood within previous 8 weeks
* Participated in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies
* Regular user of illicit drugs, or has a history of drug (including alcohol) abuse, within approximately 6 months
* Pregnant or breast-feeding, or expecting to conceive
* Interstitial lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8892 Panel A: Participants were administered MK-8892 once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 3 mg (Days 15-21), 4 mg (Days 22-28).
- MK-8892 Panel B: Participants were administered MK-8892 orally, once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 4 mg (Days 15-21), 4 mg (Days 22-28).
- MK-8892 Panel C: Participants were administered MK-8892 orally, once daily at following dose levels: 1 mg (Days 1-7), 2 mg (Days 8-14), 4 mg (Days 15-21), up to 8 mg (Days 22-28).
- Placebo (Panels A and B): Participants were administered placebo to MK-8892 once daily for 28 days.
Period: Overall Study
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C | Placebo (Panels A and B)
Started | 6 | 6 | 5 | 6
Completed | 5 | 6 | 5 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — vital sign met discontinuation criteria | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C | Placebo (Panels A and B) | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 5 | 5 | 21
  >=65 years | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 5 | 15
  Male | 2 | 4 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time-curve From Hour 0 to 24 Hours (AUC0-24hr) of MK-8892 at Day 1 and Day 28
Description: Blood samples taken at Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, and 24 hours postdose on Days 1 and 28 to determine the AUC0-24hr.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, 16, 24 hours postdose on Days 1 and 28
Population: Participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model and have data available for endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: μM*hr
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C
Number analyzed (Participants) | 6 | 6 | 5
μM*hr
  Day 1 | 0.143 [0.08 to 0.24] | 0.123 [0.017 to 0.23] | 0.192 [0.09 to 0.40]
  Day 28 | 0.863 [0.49 to 1.51] | 0.595 [0.32 to 1.11] | 1.61 [0.77 to 3.35]

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The number of participants that reported at least 1 AE was summarized.
Time Frame: Up to 42 days
Population: All participants who received at least one dose of the investigational drug
Measure: Number; unit: Participants
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C | Placebo (Panels A and B)
Number analyzed (Participants) | 6 | 6 | 5 | 6
Participants | 1 | 1 | 4 | 0

3. Primary Outcome: Number of Participants Who Had Study Drug Discontinued Due to an Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. The number of participants who had study drug discontinued due to an AE was summarized.
Time Frame: Up to 28 days
Population: All participants who received at least one dose of the investigational drug
Measure: Number; unit: Participants
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C | Placebo (Panels A and B)
Number analyzed (Participants) | 6 | 6 | 5 | 6
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: All participant that received at least 1 dose of study drug. Adverse events were summarized by randomly assigned panel.
Arm/Group | MK-8892 Panel A | MK-8892 Panel B | MK-8892 Panel C | Placebo (Panels A and B)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 4/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8892 Panel A (N=6) | MK-8892 Panel B (N=6) | MK-8892 Panel C (N=5) | Placebo (Panels A and B) (N=6)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.